CLINICAL TRIAL: NCT05431933
Title: A Multicenter, Open-label, Interventional Phase 3b Study to Evaluate the Safety, One-year Antibody Persistence, Priming Immune Responses of Three Doses of Eupolio Inj. (Inactivated Polio Vaccine (Sabin Strains)) and Immunogenicity of Two Doses of Eupolio Inj. Following Three Doses of bOPV in Infants
Brief Title: Study to Evaluate Eupolio(IPV)'s Safety, Long-term Protective Effect and Boosting Effect of One Booster Dose in the Three Primary Vaccination Plus Boosting Schedule, and Protective Effect in the Schedule With Bivalent OPV in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LG-VCCL002
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Poliomyelitis; Vaccine Reaction
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Safety group (Experimental): Three doses of Eupolio will be administered at 6, 10 and 14 weeks of age. Only safety will be evaluated for this arm.
  Interventions: Biological: Eupolio
- Immunogenicity group 1 (4 Eupolio including 1 boosting dose) (Experimental): Three doses of Eupolio will be administered at 6, 10 and 14 weeks of age, and additional single dose of Eupolio will be administered one year after the three primary vaccinations.
  Interventions: Biological: Eupolio
- Immunogenicity group 2 (3bOPV+2 Eupolio) (Experimental): bOPV will be administered at 6, 10 and 14 weeks of age, and Eupolio will be administered at 14 and 40 weeks of age.
  Interventions: Biological: Eupolio

INTERVENTIONS:
Biological: Eupolio — Inactivated Polio vaccine (Sabin strains)

SUMMARY:
Eupolio is inactivated poliovirus vaccine (IPV). Major purpose of this study is to evaluate safety of Eupolio in 2,000 infants. In addition to the safety, long-term protection after completion of the three primary vaccinations and extent of protective level after a single boosting dose of Eupolio will be evaluated.

As IPV plus bOPV vaccination schedule (3 doses of bOPV plus 2 doses of IPV in infant-toddle vaccination schedule) has been implemented in some countries, this study will also evaluate Eupolio's safety and protective effect in that schedule.

ELIGIBILITY:
Inclusion Criteria:

* Infants in stable health
* Male or female 6 to 8 weeks of age
* Signed informed consent by the infant's parent(s) or legally acceptable representative(s)

Exclusion Criteria:

* Known or suspected poliomyelitis
* Known or suspected febrile(symptom of a fever), or chronic illnesses
* Fever ≥ 38.0℃/100.4℉ within 3 days prior to study registration or intake of drug preventing fever
* Known or suspected immune disorders (abnormal activity in protective system in human body) or received immunosuppressive therapy (treatment for weaken protective system in human body)
* Previous use of blood or blood-derived products
* Previous use of polio vaccines
* Seizures (temporary abnormalities in muscle tone or movements due to abnormal activity in the brain)
* Bleeding disorders
* Household contact or intimate exposure with a confirmed case of polio
* Any history of allergy (hypersensitivity) to the components of the polio vaccine
* Participation in another interventional clinical trial simultaneously or within 30 days

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2001 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Immediate reaction | 30 minutes after each vaccination
  Any side effects that occur within 30 minutes after the vaccination
Solicited adverse event | 7 days after each vaccination
  Expected local or systemic side effects after vaccination
Unsolicited adverse event | 28 days after each vaccinations
  All unwanted or bad events after vaccination other than solicited adverse event

SECONDARY OUTCOMES:
Seroprotection rate | 4 weeks after the third vaccination, 52 weeks after the third vaccination and 7 days after the boosting vaccination in the 4 Eupolio group/ 4 weeks after the first and second vaccination in the 3bOPV+2Eupolio group
  Proportion of infants who have more than 8 protective antibody titers
Geometric mean titers of neutralizing antibody against polio antigens | 4 weeks after the third vaccination, 52 weeks after the third vaccination and 7 days after the boosting vaccination in the 4 Eupolio group / 4 weeks after the first and second vaccination in the 3bOPV+2Eupolio group
  Geometric mean titers and log2 titers for protective antibody against poliovirus type 1, 2, and 3
Priming response | 7 days after the boosting vaccination in the 4 Eupolio group
  Proportion of infants who have more than 8 protective antibody titers after boosting dose, depending on protective state before boosting dose.
Seroconversion rate | 4 weeks after the third vaccination in the 4 Eupolio group / 4 weeks after the first and second vaccination in the 3bOPV+2Eupolio group
  Proportion of infants who have more than 8 protective antibody titers after three primary vaccinations, depending on protective state before vaccination.

CONTACTS AND LOCATIONS:
Locations (10):
- Philippines (5):
  - Health Index Multispecialty and Lying-in Clinic, Cavite City
  - De La Salle Medical and Health Sciences Institue, Gov, D, Nabgybat Ave
  - University of the Philippines - Philippine General Hospital, Manila
  - Tropical Disease Foundateion, Inc., Metro Manila
  - Philippine Heart Center, Quezon City
- Thailand (5):
  - Faculty of Medicine, Chulalongkorn University, Bangkok
  - Siriraj hospital, Bangkok
  - Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Khon Kaen University, Srinagarind Hospital, Khon Kaen
  - Hatyai Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: No